CLINICAL TRIAL: NCT04112108
Title: Late (up to 12 Years) Clinical and Echocardiographic Outcomes of Percutaneous Transvenous Mitral Commissurotomy in Patients With Rheumatic Mitral Stenosis: Continuing Secondary Antibiotic Prophylaxis Does Not Protect Against Late Events
Brief Title: Late Clinical Outcomes of Percutaneous Mitral Commissurotomy in Patients With Mitral Stenosis
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Javad Kojuri, Professor, Shiraz University of Medical Sciences
Other Study IDs: 97-55318
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Mitral Valve Stenosis
Keywords: percutaneous mitral commissurotomy; follow up
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mitral stenosis post percutaneous mitral commissurotomy(PTMC): successful PTMC after follow up
  Interventions: Procedure: PTMC

INTERVENTIONS:
Procedure: PTMC — percutaneous mitral ballooning with Inoue balloon
  Other Names: mitral ballooning

SUMMARY:
In this retrospective cohort study, out of 220 patients who had undergone successful PTMC between 2006 and 2018, the clinical course of 186 patients could be successfully followed. Peri-procedural clinical and echocardiographic data were collected for these patients. Cardiac-related death, undergoing a second PTMC or mitral valve replacement (MVR) were considered adverse cardiac events in follow-up for the purpose of this study. Patients with no history of these events were contacted and asked to undergo echocardiographic imaging, in order to assess the prevalence of mitral valve restenosis, defined as mitral valve area (MVA) < 1.5 cm2 and loss of ≥50% of initial area gain

DETAILED DESCRIPTION:
This research was designed as single-technique (Inoue balloon), multicenter retrospective- prospective cohort study. The target group of this study consisted of 220 patients with symptomatic MS who had undergone PTMC at in 4 hospitals (Baqiyatallah, Namazi, Shahid-Faghihi and Kowsar) under the supervision of Baqiyatallah University of Medical Sciences and Shiraz University of Medical Sciences between April 2006 and January 2018. The demographic data of the patients were obtained from the medical records departments at each center.

The inclusion criteria for the participants were: 1) age more than 20 years at the time of PTMC; 2) immediate post-PTMC mitral valve area (IMVA) ≥1.5 cm2, or for lower values, at least 50% increase in pre-PTMC mitral valve area (MVA); 3) an initial cardiovascular event-free period of at least 6 months after the procedure.

The exclusion criteria consisted of: 1) more than 2+ mitral regurgitation (MR) immediately after the procedure; 2) immediate cardiovascular event during the hospital stay after the procedure; 3) more than mild aortic stenosis or sufficiency before PTMC; 4) history of previous PTMC or surgical mitral procedures.

The study design and steps were approved by the ethics committees at both Baqiyatallah and Shiraz University of Medical Sciences.

PTMC Technique All PTMC procedures were done with an Inoue balloon catheter by skilled interventional cardiologists via anterograde trans-septal approach in all patients. Right and left cardiac catheterization was performed before and during the procedure to assess hemodynamic changes. Optimal balloon size (in millimeters) was estimated with the height (cm)/10 + 10 formula. The balloon was inflated in a step-wise fashion from lower to higher volumes. After each inflation, changes in trans-mitral mean pressure gradient (TMPG) and the degree of mitral regurgitation (MR) were monitored. Based on interventionist's judgement and in order to achieve optimal results, balloon inflation could be continued up to 1-2 mm more than the estimated size. In the last stage, left ventriculography was conducted to assess the degree of final MR.

Echocardiography All the patient included underwent transthoracic Doppler echocardiography (TTE) in the week before PTMC by expert cardiologists with an advanced echocardiography fellowship. All general echocardiographic findings and significant mitral valve-related characteristics were reported. MVA was measured by planimetry in the short axis view, and also by pressure half-time quantification when atrial fibrillation (AF) or MR were not serious enough to interfere with its interpretation. The degree of MR was reported on a semi-quantitative scale of 0 to 4 based on Doppler color flow mapping. Mitral valve morphology was also evaluated with the standard Wilkins echocardiographic scoring system in the spectrum of 4 to 16. Pulmonary arterial pressure was estimated by measuring systolic pulmonary arterial pressure (sPAP) in mmHg based on the trans-tricuspid regurgitation jet. Other significant variables in this study were left atrial diameter in centimeters, and mean trans-mitral pressure gradient (TMPG) in mmHg.

Each patient also had one session of transesophageal echocardiography during the day before the procedure in order to rule out thrombi in the left atrium or the left atrial appendage. Another session of TTE was performed during the first day after the procedure to confirm the immediate success of PTMC, with the main focus on mitral valve-related parameters, and also to rule out acute complications such as severe MR or cardiac tamponade.

Follow-up The clinical condition of the patients was recorded as their New York Heart Association (NYHA) functional class before the procedure. Their clinical status was also followed in their inpatient and outpatient records. For the purpose of this study, the patients or their first-degree relatives were contacted by telephone in order to record the occurrence and exact timing of any adverse cardiac events, and also to reassess their current NYHA functional class status. Clinical events considered significant for the purpose of this study included: 1) cardiac-related death, 2) another session of PTMC, or 3) surgical procedure of mitral valve replacement (MVR). Patients who had been event-free until that time were asked to undergo another TTE evaluation after providing their informed consent, in order to compare the echocardiographic variables noted above with their previous records.

Statistical Analysis Continuous variables are reported as the mean ± SD. Categorical and nominal variables are shown as the number and percentage, and were pooled in some cases in order to facilitate the interpretation of the results. Initially, univariate Cox proportional hazards regression analysis was used to assess the relationship between variables and adverse cardiac events at follow-up. In the next stage, Cox multivariable regression was also performed to single out the independent variables. To evaluate the variables for the occurrence of restenosis during follow-up, uni- and multivariate logistic regression analysis was used. Receiver operating characteristic (ROC) curves were generated to determine the best cut-off point for IMVA in interpreting the results. For all analyses a p-value of 0.05 or less was considered statistically significant. All data analyses were done with IBM SPSS Statistics version 23 software.

ELIGIBILITY:
Inclusion Criteria:

* each patient with mitral stenosis undergone successful PTMC

Exclusion Criteria:

* patient refuse to took part
* inability to follow patient

Ages: 35 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: : In this retrospective cohort study, out of 220 patients who had undergone successful PTMC between 2006 and 2018, the clinical course of 186 patients could be successfully followed. Peri-procedural clinical and echocardiographic data were collected for these patients. Cardiac-related death, undergoing a second PTMC or mitral valve replacement (MVR) were considered adverse cardiac events in follow-up for the purpose of this study. Patients with no history of these events were contacted and asked to undergo echocardiographic imaging, in order to assess the prevalence of mitral valve restenosis, defined as mitral valve area (MVA) < 1.5 cm2 and loss of ≥50% of initial area gain
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
mitral stenosis | 5.6 years
  mitral valve area in echocardiographic evaluation<1.5 cm2

SECONDARY OUTCOMES:
functional class | 5.6 years
  New York heart association functional class

CONTACTS AND LOCATIONS:
Locations (1):
- Education Developmen Center, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
we have not to share data, unless all requests be evaluated by all authors

REFERENCES:
- [Derived] Dadjo Y, Moshkani Farahani M, Nowshad R, Sadeghi Ghahrodi M, Moaref A, Kojuri J. Mid-term (up to 12 years) clinical and echocardiographic outcomes of percutaneous transvenous mitral commissurotomy in patients with rheumatic mitral stenosis. BMC Cardiovasc Disord. 2021 Jul 28;21(1):355. doi: 10.1186/s12872-021-02175-3. PMID 34320949